CLINICAL TRIAL: NCT05520138
Title: A Real-World Comparison of Clinical Outcomes in Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer (mCRPC) Patients Who Initiated Enzalutamide vs. Abiraterone Acetate (Abiraterone) in the 100% Medicare Fee-For-Service (FFS) Data (2009-2020)
Brief Title: Enzalutamide vs. Abiraterone in Chemotherapy-naïve Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3431046; Enza vs Abi rwOS in Medicare (Other: Alias Study Number)
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: metastatic castration-resistant prostate cancer; mCRPC; enzalutamide; abiraterone; overall survival; OS; treatment duration
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — enzalutamide; Abiraterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Enzalutamide cohort: Patients with mCRPC initiating enzalutamide
  Interventions: Drug: Enzalutamide
- Abiraterone cohort: Patients with mCRPC initiating abiraterone
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Enzalutamide — As provided in real-world setting
  Other Names: Xtandi
  Groups: Enzalutamide cohort
Drug: Abiraterone acetate — As provided in real-world setting
  Other Names: Yonsa, Zytiga
  Groups: Abiraterone cohort

SUMMARY:
This study will be a retrospective data analysis to compare outcomes between patients with chemotherapy-naïve metastatic castration-resistant prostate cancer (mCRPC) who initiated enzalutamide and those who initiated abiraterone using the 100% Fee-For-Service Medicare claims data. The study will address the following objectives:

Primary objective: To compare overall survival (OS) in patients with chemotherapy-naïve mCRPC who initiated enzalutamide vs. abiraterone

Secondary objectives:

* To compare OS in patients with chemotherapy-naïve mCRPC who received only enzalutamide without any subsequent therapy vs. abiraterone without any subsequent therapy
* To compare treatment duration and time to subsequent therapy in chemotherapy-naïve mCRPC patients initiating enzalutamide vs. abiraterone

ELIGIBILITY:
Inclusion Criteria:

* Male with ≥ 1 diagnosis claim for prostate cancer
* Have documented secondary metastasis code on or after the initial prostate cancer diagnosis
* Have initiated enzalutamide or abiraterone within 90 days prior to the metastasis date or on or after the metastasis date. The initiation date of enzalutamide or abiraterone will be defined as the index date.
* Have evidence of surgical or medical castration before the index date
* At least 18 years old at the index date
* Continuous eligibility for ≥ 12 months prior to the index date

Exclusion Criteria:

* Received chemotherapy, novel hormonal therapy, radium-223, or immunotherapy prior to the index date
* Had a prior history of other cancers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chemotherapy-naïve mCRPC (aged ≥18 years) who initiated enzalutamide or abiraterone and met eligibility criteria will be included in the study. Patients will be identified from the 100% Fee-For-Service Medicare claims data.
Sampling Method: Non-Probability Sample
Enrollment: 5506 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3431046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants- with chemotherapy naive metastatic castration-resistant prostate cancer (mCRPC), who initiated abiraterone or enzalutamide during the index period of 10 September 2014 to 31 May 2017 (approximately 33 months)- were included in this study. Data was retrieved from 100% Medicare Fee-For-Service (FFS). Retrospective data extracted and evaluated from study start date and until study completion (approximately 10 months) of this retrospective observational study.
Groups:
- Abiraterone: Participants with mCRPC who initiated abiraterone during the index period in real-world setting and whose data were observed in the study, were included in this reporting group.
- Enzalutamide: Participants with mCRPC who initiated enzalutamide during the index period in real-world setting and whose data were observed in the study, were included in this reporting group.
Period: Overall Study
Arm/Group | Abiraterone | Enzalutamide
Started | 2911 | 2595
Completed | 2911 | 2595
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone | Enzalutamide | Total
Number analyzed (Participants) | 2911 | 2595 | 5506
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.4 (7.9) | 78.6 (8.2) | 78.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2911 | 2595 | 5506
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 364 | 336 | 700
  White, non-Hispanic | 2273 | 2012 | 4285
  Hispanic | 148 | 134 | 282
  Unknown or Others | 126 | 113 | 239

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS): Inverse Probability Treatment Weighting (IPTW)
Description: OS (time to death) was defined as the time from the initiation of enzalutamide or abiraterone (i.e., index date) to the date of death. Participants who did not die were censored at their last available follow-up, which was defined as the earlier of disenrollment from Medicare or end of data availability. Kaplan-Meier method was used for analysis.
Time Frame: From index date to date of death or censoring date, whichever occurred first (from 10-Sep-2014 to 31-Dec-2020, approximately 76 months); retrospective data extracted and evaluated from study start date and until study completion (approximately 10 months)
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, ''Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure after adjusting for baseline confounders (demographics, clinical characteristics, prior treatments, comorbidities, medical resource use) using IPTW. Hence, numbers are different here from those presented in participant and baseline section.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone | Enzalutamide
Number analyzed (Participants) | 2912 | 2591
Months | 20.6 [19.7 to 21.4] | 22.5 [21.2 to 23.8]
Statistical Analysis 1: Comparison: Abiraterone vs Enzalutamide; Test type: Superiority — With a 2-sided Type I of 0.05 significance; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [1.04 to 1.16] — A weighted Cox proportional hazard model with an independent variable for treatment group were fitted, using a robust variance estimator

2. Secondary Outcome: OS Among Participants Without Any Subsequent Therapy: IPTW
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone | Enzalutamide
Number analyzed (Participants) | 1168 | 1075
Months | 10.6 [9.6 to 11.7] | 13.6 [12.4 to 15.1]
Statistical Analysis 1: Comparison: Abiraterone vs Enzalutamide; Test type: Superiority — With a 2-sided Type I of 0.05 significance; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [1.06 to 1.27] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Treatment Duration: IPTW
Description: Treatment duration of the index treatment was defined as the time from the initiation of enzalutamide or abiraterone (i.e., index date) to the discontinuation date. Discontinuation was defined as the earliest of 1) death, 2) last observed administration plus day of supply associated with last administration, or 3) day before the start of next line of therapy. Death, a gap of 90 days or more after the last observed prescription date + day of supply, and initiation of next line of therapy was considered as discontinuation events. Participants who did not discontinue were censored at their last available follow-up, which was defined as the earlier of disenrollment from Medicare or end of data availability.
Time Frame: From index date to date of discontinuation event or censoring date, whichever occurred first(from 10-Sep-2014 to 31-Dec-2020, approximately 76months); retrospective data extracted and evaluated from start date and until completion(approximately 10months)
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here ''Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure after adjusting for baseline confounders (demographics, clinical characteristics, prior treatments, comorbidities, medical resource use) using IPTW. Hence, numbers are different here from those presented in participant and baseline section.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone | Enzalutamide
Number analyzed (Participants) | 2912 | 2591
Months | 6.7 [6.3 to 7.0] | 7.4 [7.0 to 7.9]
Statistical Analysis 1: Comparison: Abiraterone vs Enzalutamide; Test type: Other; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.99 to 1.10] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Subsequent Therapy: IPTW
Description: Time to subsequent therapy was defined as the time from the initiation of enzalutamide or abiraterone (i.e., index date) to the start of next line of therapy. Participants who did not start a new line of therapy were censored at their last available follow-up, which was defined as the earliest of 1) death, 2) disenrollment from Medicare, and 3) end of data availability.
Time Frame: From index date to start of next line of therapy (from 10-Sep-2014 to 31-Dec-2020, approximately 76 months); retrospective data extracted and evaluated from study start date and until study completion (approximately 10 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone | Enzalutamide
Number analyzed (Participants) | 2912 | 2591
Months | 14.5 [13.4 to 15.4] | 16.7 [15.9 to 17.8]
Statistical Analysis 1: Comparison: Abiraterone vs Enzalutamide; Test type: Other; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [1.06 to 1.22] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: For mortality: from 10-Sep-2014 to 31-Dec-2020 (approximately 76 months); retrospective data extracted and evaluated from study start date and until study completion (approximately 10 months) of this retrospective observational study; Adverse events: Not applicable as adverse events were not planned to be collected during the study
Description: From data source, individual participant data were not retrieved or validated. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) cannot be met. Hence, adverse events were not collected and reported.
Arm/Group | Abiraterone | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 2523/2911 | 2176/2595
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT05520138/Prot_SAP_000.pdf